CLINICAL TRIAL: NCT01548586
Title: Modulation de l'excitabilité Des Aires Corticales Motrices Primaires Correspondant Aux hémi Diaphragmes à l'Aide de la tDCS (Transcranial Direct Current Stimulation)
Brief Title: Effect of Transcranial Direct Current Stimulation (tDCS) on the Excitability of the Diaphragmatic Primary Motor Cortex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C10-52; 2011-A00508-33 (Registry Identifier: Numéro IDRCB)
Record Dates: First submitted 2012-01-23; First posted 2012-03-08 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2021-08

CONDITIONS: Excitability of Diaphragmatic Primary Motor Cortex
Keywords: tDCS; Diaphragm; Cortical Excitability; MEPs; TMS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Anodal tDCS (Active Comparator)
  Interventions: Device: Eldith DC stimulator ( Magstim Company Ltd. UK)
- Cathodal tDCS (Active Comparator)
  Interventions: Device: Eldith DC stimulator ( Magstim Company Ltd. UK)
- Placebo type tDCS (Placebo Comparator)
  Interventions: Device: Eldith DC stimulator ( Magstim Company Ltd. UK)

INTERVENTIONS:
Device: Eldith DC stimulator ( Magstim Company Ltd. UK) — Anodal tDCS: Intensity of 2 mA , during 10 min Cathodal tDCS: Intensity of 2 mA , during 10 min Placebo type tDCS: Intensity of 0 mA during 10 min
  Other Names: Magstim 200 TMS(Magstim Company Ltd.UK)

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non invasive, painless, harmless way to modulate cerebral cortex excitability. It was shown that anodal stimulation increases cortical excitability and the cathodal one decreases it (Nitsche and Paulus, 2000; Lang et al. 2004). To date, there is no data in the literature regarding the effect of tDCS on the corticodiaphragmatic pathways. This preliminary study aims to test and validate the modulating effect of tDCS on the excitability of the primary motor cortex dedicated to the hemi-diaphragms in a sample of healthy subjects, as a prelude to further large studies in patients with paretic hemi-diaphragms. Diaphragmatic motor evoked potentials will be assessed before and after applications of three different modalities of tDCS (anodal, cathodal and placebo).

DETAILED DESCRIPTION:
We therefore expect to observe a significant increase of the mean values of the right hemidiaphragm's MEP's amplitudes after application of anodal tDCS compared to the baseline MEP obtained before this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Right handed,
* Healthy male volunteers
* Aged ≥ 18 and ≤ 35 years
* No history of neurological or respiratory disease
* BMI (body mass index < 30)

Exclusion Criteria:

* Female sex
* Vulnerable people as defined in the provisions relating to biomedical researches and described in the Code of Public Health.
* Recent or ongoing use of antibiotic drugs, antidepressants or psychotropic drugs.
* Recent hospitalization (within 3 months).
* No affiliation to a social security system.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in the right side hemi-diaphragm's motor evoked potentials (MEPs) before and after applications of three different modalities of tDCS (anodal, cathodal and placebo) upon the left primary motor cortex. | Baseline MEPs (before tDCS), Post 0 MEPs (immediately after tDCS) and Post 10 MEPs (10 min after tDCS).
  The facilitating effect of tDCS in Anodal stimulation mode (a-tDCS) on the excitability of the left diaphragmatic primary motor cortex would result in a significant increase of the amplitude of the right hemidiaphragm motor evoked potentials (MEPs) (obtained by Transcranial magnetic motor stimulation of the left diaphragmatic primary) after this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric AZABOU, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Fréderic LOFASO, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpitaux Universitaires Paris Ile de France Ouest - Hôpital Raymond poincaré, Garches, Île-de-France Region, France

REFERENCES:
- [Background] Azabou E, Roche N, Sharshar T, Bussel B, Lofaso F, Petitjean M. Transcranial direct-current stimulation reduced the excitability of diaphragmatic corticospinal pathways whatever the polarity used. Respir Physiol Neurobiol. 2013 Oct 1;189(1):183-7. doi: 10.1016/j.resp.2013.07.024. Epub 2013 Aug 7. PMID 23933029
- [Background] Hummel F, Celnik P, Giraux P, Floel A, Wu WH, Gerloff C, Cohen LG. Effects of non-invasive cortical stimulation on skilled motor function in chronic stroke. Brain. 2005 Mar;128(Pt 3):490-9. doi: 10.1093/brain/awh369. Epub 2005 Jan 5. PMID 15634731
- [Background] Madhavan S, Stinear JW. Focal and bi-directional modulation of lower limb motor cortex using anodal transcranial direct current stimulation. Brain Stimul. 2010 Jan;3(1):42. doi: 10.1016/j.brs.2009.06.005. PMID 20161639
- [Background] Nitsche MA, Paulus W. Transcranial direct current stimulation--update 2011. Restor Neurol Neurosci. 2011;29(6):463-92. doi: 10.3233/RNN-2011-0618. PMID 22085959
- [Background] Nitsche MA, Seeber A, Frommann K, Klein CC, Rochford C, Nitsche MS, Fricke K, Liebetanz D, Lang N, Antal A, Paulus W, Tergau F. Modulating parameters of excitability during and after transcranial direct current stimulation of the human motor cortex. J Physiol. 2005 Oct 1;568(Pt 1):291-303. doi: 10.1113/jphysiol.2005.092429. Epub 2005 Jul 7. PMID 16002441
- [Background] Nitsche MA, Paulus W. Sustained excitability elevations induced by transcranial DC motor cortex stimulation in humans. Neurology. 2001 Nov 27;57(10):1899-901. doi: 10.1212/wnl.57.10.1899. PMID 11723286
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Roche N, Lackmy A, Achache V, Bussel B, Katz R. Impact of transcranial direct current stimulation on spinal network excitability in humans. J Physiol. 2009 Dec 1;587(Pt 23):5653-64. doi: 10.1113/jphysiol.2009.177550. Epub 2009 Oct 5. PMID 19805746
- [Background] Sharshar T, Hopkinson NS, Jonville S, Prigent H, Carlier R, Dayer MJ, Swallow EB, Lofaso F, Moxham J, Polkey MI. Demonstration of a second rapidly conducting cortico-diaphragmatic pathway in humans. J Physiol. 2004 Nov 1;560(Pt 3):897-908. doi: 10.1113/jphysiol.2004.061150. Epub 2004 Jul 22. PMID 15272049
- [Background] Similowski T, Catala M, Rancurel G, Derenne JP. Impairment of central motor conduction to the diaphragm in stroke. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):436-41. doi: 10.1164/ajrccm.154.2.8756819.
- See also: This paper reports results of this study — https://uvsq.hal.science/hal-02614100v1/document
- See also: This paper reports results of this study — https://uvsq.hal.science/hal-01911136/document